CLINICAL TRIAL: NCT00035854
Title: Linezolid IV/PO for the Treatment of Vancomycin-Resistant Enterococcus Infections in Children
Brief Title: New Antibiotic to Treat Pediatric Patients With Infections Due to a Specific Bacteria (Vancomycin-Resistant Enterococcus)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12600082VRE; A5951062
Record Dates: First submitted 2002-05-06; First posted 2002-05-07 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Bacterial Infections
Keywords: Pharmacia; Drug Resistance, Microbial
MeSH Terms: conditions — Bacterial Infections | interventions — Linezolid

INTERVENTIONS:
Drug: Zyvox® / Linezolid

SUMMARY:
This study will treat pediatric patients who have infections that are due to a specific bacteria (Vancomycin-Resistant Enterococcus)

ELIGIBILITY:
Other specific inclusion/exclusion criteria may apply. In order to determine eligibility, further examination by the investigator is necessary.

Inclusion Criteria:

* Hospitalized/chronic care pediatric patients (birth through 17 years)
* Known infections due to vancomycin-resistant enterococcus species, including diagnosis of hospital-acquired pneumonia, complicated skin and skin structure infections, catheter-related bacteremia, bacteremia of unidentified source, and other infections
* Requires a minimum of 3 days of IV medication
* Patients with mixed infections due to VRE & gram negative bacteria are allowed to enroll in the study. For most of the infections, 2 or more of additional symptoms are required.

Exclusion Criteria:

* Potentially effective concomitant antibiotic
* A high surgical cure rate
* Medical conditions which would preclude clinical evaluation or require treatment of longer duration than 28 days
* 24 hours of antibiotic treatment within 48 hours of study entry (unless pre-approved)
* Having an infected device that could not be removed

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2002-02; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Investigator's and sponsor's evaluation of patient clinical outcome.

SECONDARY OUTCOMES:
Pathogen eradication rates, changes in clinical signs and symptoms, body temperature, WBC count, lesion size (for SSSIs) and chest radiograph findings(for HAP).

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Research Center, Long Beach, California
  - Research Center, Los Angeles, California
  - Research Center, Hartford, Connecticut
  - Research Center, Washington D.C., District of Columbia
  - Research Center, Gainesville, Florida
  - Research Center, Atlanta, Georgia
  - Research Center, Chicago, Illinois
  - Research Center, Park Ridge, Illinois
  - Research Center, Louisville, Kentucky
  - Research Center, Baltimore, Maryland
  - Research Center, Boston, Massachusetts
  - Research Center, Detroit, Michigan
  - Research Center, Camden, New Jersey
  - Research Center, New York, New York
  - Research Center, Cleveland, Ohio
  - Research Center, Danville, Pennsylvania
  - Research Center, Philadelphia, Pennsylvania
  - Research Center, Austin, Texas